CLINICAL TRIAL: NCT01381315
Title: ARM: Axillary Reverse Mapping
Brief Title: Axillary Reverse Mapping
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11737
Record Dates: First submitted 2011-06-09; First posted 2011-06-27 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: Sentinel lymph node biopsy; Axillary lymph node dissection; Prevention of lymphedema
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sentinel lymph node biopsy (Other): During surgery, 1.0 mCi of technetium-99m sulfur colloid will be injected into sub-dermal subareolar aspect of the affected breast. The KUMC Nuclear Medicine Department will be responsible for performing the injection of the isotope and dilution of the isotope using saline to a final volume of 4.0 ml or less.
  Interventions: Procedure: Injection of isotope
- Axillary lymph node biopsy (Other)
  Interventions: Procedure: Axillary lymph node dissection

INTERVENTIONS:
Procedure: Injection of isotope — On the day of surgery, if the radioactive SLN cannot be located using the gamma probe prior to incision, lymphazurin or methylene blue dye will be used in the breast in the subareolar plexus at the discretion of the surgeon for assistance in identifying the sentinel nodes. This contingency, expected to occur <3% of the time, will be used since locating the SLN for staging is of greater importance than the study. If radioactive isotope is sufficient to identify the sentinel node draining from the breast, then the blue dye will be injected dermally in the upper inner arm along the bicipital groove of the ipsilateral arm in order to locate the draining lymphatics from the arm. No more than 5cc of blue dye will be injected in any of the above mentioned scenarios.
  Arms: Sentinel lymph node biopsy
Procedure: Axillary lymph node dissection — The one-year lymphedema rate among subjects undergoing axillary lymph node dissection with or without sentinel lymph node biopsy is ≥ 0.13. With our sample size of 58 subjects undergoing ALND, we will reject that hypothesis in favor of the alternative-that the lymphedema rate is <0.13 for subjects undergoing ALND-if lymphedema is confirmed in three or fewer (ie, 0, 1, 2, or 3) subjects.
  Arms: Axillary lymph node biopsy

SUMMARY:
It has been hypothesized that the proximity of the anatomic locations of the arm lymphatic drainage system to the breast lymphatic system in the axilla put the arm lymphatics at risk for disruption during a sentinel lymph node biopsy (SLNB) and/or axillary lymph node dissection (ALND). Therefore, mapping the drainage of the arm in addition to the drainage of the breast during the procedure would potentially decrease the incidence of arm lymphatic disruption and subsequent development of lymphedema while providing adequate axillary breast nodes needed for staging.

DETAILED DESCRIPTION:
Patients will receive an injection of 1.0 mCi of technetium-99m sulfur colloid that will be injected into the sub-dermal subareolar aspect of the affected breast.

On the day of surgery, if the radioactive SLN cannot be located using the gamma probe prior to incision, lymphazurin or methylene blue dye will be used in the breast in the subareolar plexus at the discretion of the surgeon for assistance in identifying the sentinel nodes. This contingency, expected to occur < 3% of the time, will be used since locating the SLN for staging is of greater importance than the study. If radioactive isotope is sufficient to identify the sentinel node draining from the breast, then the blue dye will be injected dermally in the upper inner arm along the bicipital groove of the ipsilateral arm in order to locate the draining lymphatics from the arm. No more than 5cc of blue dye will be injected in any of the above mentioned scenarios. The site of all injections (radioactivity and/or blue dye) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 100 years old
* Not pregnant or breastfeeding
* Diagnosis of breast cancer requiring LN evaluation for ipsilateral or contralateral breast or prophylactic mastectomy
* Willing participation after obtaining informed consent

Exclusion Criteria:

* < 18 or > 100 years of age
* Pregnant or breastfeeding
* Blue dye allergy
* Cosmetic allergy
* History of primary lymphedema
* Prior breast augmentation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2009-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Assess lymphedema rates | Four Years
  The primary objective of this study is to assess and test the lymphedema rates six times at the following intervals: Pre-surgery - baseline, at 6 months, and yearly for 4 years. Since the historical control rates are different (5% for SLNB only and 13% for ALND with or without SLNB) two tests will be performed.

SECONDARY OUTCOMES:
Identification of breast sentinal lymph node and arm lymphatics | at time of surgery
  Successful identification (localization) of breast sentinel lymph node and arm lymphatics
Characterization of location | at time of surgery
  Characterization of location (typical versus variant) of arm lymphatics
Protection of the arm | at time of surgery
  Successful protection of the arm lymphatics during sentinel lymph node biopsy and/or axillary lymph node dissection
Occurrence of crossover | at time of surgery
  Occurrence of crossover (i.e., co-localization) between hot breast sentinel lymph node and blue arm lymphatics

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Wagner, DO, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States